CLINICAL TRIAL: NCT07008508
Title: Incidence of Venous Thromboembolism and Cardiovascular Events in Breast Cancer Patients Undergoing Cyclin-dependent Kinase 4/6 Inhibitors: The Breast Cancer Associated Vascular Events During Cyclin-dependent Kinase 4/6 Inhibitors Therapy (BRAVE-Cyclin) Study
Acronym: BRAVE-Cyclin
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Pola Roberto, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ID7674
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: venous thromboembolism; breast cancer; Cyclin-dependent Kinase 4/6 Inhibitors; CDK 4/6 Inhibitors; cardiovascular disease; Palbociclib; Ribociclib; Abemaciclib
MeSH Terms: conditions — Breast Neoplasms; Venous Thromboembolism; Cardiovascular Diseases | interventions — palbociclib; abemaciclib; ribociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Cyclin-dependent Kinase 4/6 Inhibitor — Planned new line of Cyclin-dependent Kinase 4/6 Inhibitor
  Other Names: Palbociclib; Abemaciclib; Ribociclib

SUMMARY:
"Incidence of Venous Thromboembolism and Cardiovascular Events in Patients with Breast Cancer Treated with Cyclin-Dependent Kinase Inhibitors 4/6, the BRAVE-Cyclin Study" is national, single-center, observational, prospective cohort study, conducted at Fondazione Policlinico Universitario A. Gemelli IRCCS.

According to recent evidence, patients with advanced or metastatic breast cancer receiving cyclin-dependent kinase (CDK) 4/6 inhibitors - ribociclib, palbociclib, and abemaciclib - may have an increased risk of arterial or venous thrombosis.

Currently, there are no validated tools to stratify breast cancer patients receiving CDK 4/6 inhibitors according to their thromboembolic or cardiovascular risk.

The prospective BRAVE-Cyclin study aims to evaluate the incidence of venous thromboembolism, major cardiovascular events, and major adverse peripheral vascular events in breast cancer patients receiving CDK 4/6 inhibitors.

The objective is to identify the main determinants of thromboembolic and cardiovascular risk, thus improving risk stratification and management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Female sex;
* Diagnosis of advanced or metastatic breast cancer.
* Indication for therapy with Cyclin-dependent Kinase 4/6 Inhibitor, as clinical practice;
* Age of 18 years or older;
* Signing Informed Consent.

Exclusion Criteria:

• Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of subsequent patients prospectively enrolled in case of indication of systemic antineoplastic treatment with CDK 4/6 Inhibitor for advanced breast cancer. Patients will be recruited in the setting of the Gynecologic Oncology Day Hospital and evaluated by the U.O.S.D Percorso Trombosi of the Agostino Gemelli University Polyclinic Foundation I.R.C.C.S. in Rome.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2032-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
• Incidence rate of vascular events | From enrollment to the end of 60 months follow-up
  Vascular events are defined as episodes of Venous Thromboembolism (VTE) in usual or unusual site, Major Adverse Cardiovascular Events (MACE), and/or Major Adverse Limbs Events (MALE)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No